CLINICAL TRIAL: NCT06101056
Title: Code of Respect (X-CoRe): a Randomized Controlled Trial of a Multi-level Sexual Assault and Sexual Harassment Prevention Intervention for Active Duty Airmen
Brief Title: Code of Respect (X-CoRe): Trial of a Multi-level Sexual Assault and Sexual Harassment Prevention Intervention for Active Duty Airmen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Belinda Hernandez, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0619
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sexual Assault; Sexual Harassment
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Intervention Model Description: Participants will be cluster-randomized at the level of the squadron to one of two conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Code of Respect (X-CoRe) Multi-Level Sexual Assault (SA) and Harassment (SH) Prevention Program (Experimental)
  Interventions: Behavioral: Junior Enlisted Component; Behavioral: Leadership Component; Behavioral: Social Marketing Campaign
- Control Condition (Other)
  Interventions: Behavioral: Leadership Component; Behavioral: Social Marketing Campaign

INTERVENTIONS:
Behavioral: Junior Enlisted Component — Junior Enlisted Airmen (E4 and below) will complete 10 online modules designed to train them on recognizing SH and SA, healthy and unhealthy relationships, and situations that may increase risk for SH and SA. Participants will adopt and practice a lifestyle paradigm of select-detect-protect, in which service members select their personal rule to have only healthy (non-abusive) relationships with their peers and romantic partners, detect signs and situations that might threaten their rules, and protect their rules using communication, management, and avoidance skills. They will be instructed to adopt a zero-tolerance approach to SH and SA and will receive skills training related to communication and conflict resolution for healthy relationships, reduction of SH and SA perpetration, consent communication, reporting incidents of SH and SA, and bystander intervention. Participants who have experienced SH or SA are encouraged to use the "Get Help Now" feature to access support 24/7.
  Arms: Code of Respect (X-CoRe) Multi-Level Sexual Assault (SA) and Harassment (SH) Prevention Program
Behavioral: Leadership Component — Mid- and advanced-level leaders (E5 and above) will complete 10 online modules designed to train them to recognize forms of SH and SA, how to respond to an incident of SH or SA, and how to create a safe work environment free of SH and SA. Leaders will also adopt and practice the paradigm select-detect-protect. Leaders will select their personal rule to enforce a healthy work environment (free of SH and SA), detect signs and situations that might threaten their rule (e.g., displaying inappropriate pictures on the computer), and protect their rules using communication and management skills. Leaders will also be given background material on SH and SA in the military (e.g., extent of the problem, DoD definitions, and policies) and installation resources for reporting incidents. As with the Junior Enlisted component, Leaders who may have experienced SH or SA are encouraged to use our "Get Help Now" feature to access support 24/7.
Behavioral: Social Marketing Campaign — All participating Airmen (including Junior Enlisted Airmen and Leaders) will be exposed to X-CoRe's social marketing campaign, which includes posters, flyers, postcards, and digital content for social media. Messages are designed to increase awareness of consent and foster Wing-wide norms that are supportive of healthy relationships. Resources for Service members to receive support if they have experienced SH or SA will also be provided through the social marketing materials. Social marketing materials, such as posters, will be distributed at "hot spots" for SA (e.g., dorms).

SUMMARY:
The purpose of this study is to examine the efficacy of Code of Respect (X-CoRe) multi-level sexual assault (SA) and harassment (SH) prevention program in improving psychosocial determinants (e.g., knowledge, skills, self-efficacy, attitudes) related to respectful/disrespectful relationships, to examine the efficacy of X-CoRe in reducing SA and sexual harassment SH victimization and to examine the efficacy of X-CoRe increasing bystander behavior and improving unit cohesion and mission readiness by decreasing secondary risk and harmful behaviors (e.g., alcohol misuse, intimate partner violence, suicide ideation). The study will be conducted at at Joint Base McGuire Dix-Lakehurst (JBMDL) located in Burlington County, New Jersey, and participants will be cluster-randomized at the level of the squadron to one of two conditions: the X-CoRe program or a control condition.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty, stationed at JBMDL
* assigned to one of the 26 Air Force squadrons within the three Air Force Wings at JBMDL (87 Air Base Wing (ABW), 305 Air Mobility Wing (ABM), and 621 Contingency Response Wing (CRW))
* English speaking
* access to an electronic device with internet capabilities

Exclusion Criteria:

* being in service branches other than Air Force (e.g., Army or Navy)
* Airmen not ranked E1-E4 at JBMDL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in SA victimization as assessed by the Sexual Experiences Survey | baseline,6 months follow up, 12 months follow up
  This is a 10 item questionnaire and each is scored on a 4 point scale from 0-3 or more higher number indicating worse outcome
Change in SH victimization as assessed by the (Sexual Experience Questionnaire (SEQ-DoD) | baseline, 6 months follow up, 12 months follow up
  This is a 23 item questionnaire and each is scored on a 5 point scale from 0, 1-2,3-5,6-9 or more, higher number indicating worse

SECONDARY OUTCOMES:
Change in knowledge of Sexual Harassment and Assault as assessed by the Knowledge of Sexual Harassment and Assault Scale | baseline,6 months follow up, 12 months follow up
  This is a 6 item questionnaire and each question is answered as true or false
Change in Rape Myth Acceptance as assessed by the Illinois Rape Myth Acceptance Scale -Short Form | baseline,6 months follow up, 12 months follow up
  This is a 20 item questionnaire and each is scored on a 7 point scale from not at all agree-very much agree a higher number indicating worse outcome
Change in Gender Role Beliefs as assessed by the Hypergender Ideology Scale -Short Form | baseline,6 months follow up, 12 months follow up
  This is a 19 item questionnaire and each is scored on a 6 point scale from strongly disagree to strongly agree, higher number indicating worse outcome
Change in attitudes towards Sexual Harassment as assessed by the Sexual Harassment Attitude Scale | baseline,6 months follow up, 12 months follow up
  This is a 17 item questionnaire and each is scored on a 5 point scale from strongly disagree-strongly agree, higher number indicating worse outcome
Change in Attitudes towards Relationship Violence as assessed by the Acceptance of Couple Violence Scale | baseline,6 months follow up, 12 months follow up
  This is a 17 item questionnaire and each is scored on a 4 point scale from strongly disagree-strongly agree , higher number indicating worse outcome
Change in Relationships Skills Self-Efficacy as assessed by the Interpersonal competence Questionnaire - Negative assertion subscale | baseline,6 months follow up, 12 months follow up
  This is an 8 item questionnaire and each is scored on a 5 point scale from I am poor at this-I am extremely good at this, lower number indicating worse outcome
Change in Attitudes towards Preventing Sexual Harassment and Assault as assessed by the Attitudes Toward Preventing Dating Violence Subscale | baseline,6 months follow up, 12 months follow up
  This is a 3 item questionnaire and each is scored on a 4 point scale from strongly disagree to strongly agree, higher number indicating better outcome
Change in Attitudes towards Cyberbullying as assessed by the Harmful Cyberbullying Attitudes Scale | baseline,6 months follow up, 12 months follow up
  This is a 5 item questionnaire and each is scored on a 5 point scale from strongly disagree to strongly agree
  , higher number indicating worse outcome
Change in attitudes towards Alcohol Use as assessed by the Drinking Values Scale | baseline,6 months follow up, 12 months follow up
  This is a 10 item questionnaire and each is scored on a 5 point scale from strongly disagree to strongly agree, higher number indicating worse outcome
Change in Bystander Self-Efficacy as assessed by the Bystander Efficacy Scale | baseline,6 months follow up, 12 months follow up
  This is an 18 item questionnaire and each is scored from 0(can't do) to 100(very certain) higher number indicating better outcome
Change in Barriers to Sexual Assault Intervention as assessed by the Barriers to Sexual Assault Bystander Intervention Scale | baseline,6 months follow up, 12 months follow up
  This is a 23 item questionnaire and each is scored on a 7 point scale from strongly disagree-strongly agree a higher number indicating worse outcome
Change in Conflict Communication Skills as assessed by the Conflict Communication Scale - Confrontation Subscale | baseline,6 months follow up, 12 months follow up
  This is a 15 item questionnaire and each is scored on a 6 point scale from strongly disagree-strongly agree a higher number indicating worse outcome
Change in Bystander Behavior as assessed by the Bystander Behavior Scale - Risky Situations and Party Safety Subscale | baseline,6 months follow up, 12 months follow up
  This is a 25 item questionnaire and each is scored on a 4 point scale categorically from 0, 1, 2,3 or more times a higher number indicating better outcome
Change in Horizontal Unit Cohesion as assessed by the Horizontal Cohesion Scale | baseline,6 months follow up, 12 months follow up
  This is a 6 item questionnaire and each is scored on a 5 point scale from strongly disagree-strongly agree a higher number indicating better outcome
Change in Vertical Unit Cohesion as assessed by the Vertical cohesion Scale | baseline,6 months follow up, 12 months follow up
  This is a11 item questionnaire and each is scored on a 5 point scale from strongly disagree-strongly agree a higher number indicating better outcome
Change in Intimate Partner Violence as assessed by the Composite Abuse Scale (Revised) - Short Form | baseline,6 months follow up, 12 months follow up
  This is a 15 item questionnaire and each is scored on a 5 point scale from not in the past 12 months to daily/almost daily a higher number indicating worse outcome
Change in Alcohol Use as assessed by the Alcohol 30-day Quantity and Frequency | baseline,6 months follow up, 12 months follow up
  Participants are asked the following two questions: one regarding the frequency of consumption (number of days), and a second regarding the usual quantity of consumption (number of drinks) on drinking days, higher number indicating more alcohol use
Change in Suicide Ideation as assessed by the Columbia -Suicide Severity Rating Scale - Severity of Suicidal Ideation Subscale | baseline,6 months follow up, 12 months follow up
  This is a 5 item questionnaire and each is scored on a 5 point scale from wish to be dead-suicidal intent with plan a higher number indicating worse outcome
Change in Anxiety as assessed by the Generalized Anxiety Disorder Screener | baseline,6 months follow up, 12 months follow up
  This is a 7 item questionnaire and each is scored on a 4 point scale from not at all-nearly every day a higher number indicating worse outcome
Change in Depression as assessed by the Patient Health Questionnaire 9 (PHQ-9) | baseline,6 months follow up, 12 months follow up
  This is a 9 item questionnaire and each is scored on a 4 point scale from not at all-nearly every day a higher number indicating worse outcome
Change in PTSD as assessed by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Cross Cutting Symptom Measure | baseline,6 months follow up, 12 months follow up
  This is a 23 item questionnaire and each is scored on a 5 point scale from not at all-nearly every day a higher number indicating worse outcome
Change in Overall Health Functioning as assessed by the World Health Organization Disability Assessment Schedule (WHODAS) 2.0) - Short Form | baseline,6 months follow up, 12 months follow up
  This is a 12 item questionnaire and each is scored on a 5 point scale from none-extreme or cannot do a higher number indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Hernandez, PhD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No